CLINICAL TRIAL: NCT03840044
Title: The Effect of Physical Exercise in a Cold Air Environment on Normal Volunteers and Asthmatic Patients
Acronym: ALASCAIR1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Tatjana Decaesteker, Co-Principal Investigator, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: s61661
Record Dates: First submitted 2019-01-23; First posted 2019-02-15 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Asthma, Exercise-Induced
Keywords: Asthma; Exercise; Cold air exposure
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Healthy volunteers will be compared with asthmatic subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Other): Healthy volunteers will perform the same protocol as foreseen for asthmatic patients. Both will perform the cold air exercise test with pre -and post-exposure evaluation of on FEV1, respiratory symptoms, functional airway integrity, local and systemic inflammation and on the airway microbiome.
  Interventions: Other: Cold air exercise test
- Asthmatic subjects (Other): Asthmatic patients will perform the same protocol as foreseen for healthy volunteers. They will perform the cold air exercise test with pre -and post-exposure evaluation of on FEV1, respiratory symptoms, functional airway integrity, local and systemic inflammation and on the airway microbiome.
  Interventions: Other: Cold air exercise test

INTERVENTIONS:
Other: Cold air exercise test — Subjects will perform a submaximal 90 minutes exercise test in a controlled cold air environment (-5°C, 60% relative humidity) in a climate chamber with evaluation pre§/during*/post§ of heart rate (HR)§* and blood pressure (BP)§*, spirometry§*, PNIF§, FeNO§, electrocardiogram (ECG)§*, body & exhaled air temperature§*, capsaicin cough threshold test§, histamine bronchial challenge test§, and sampling of nasal fluid§, induced sputum§, and venous blood§.

SUMMARY:
The purpose of the study is to compare airway physiologic reactions to physical exercise in a cold air environment (-5°C, 60% relative humidity) between normal volunteers and subjects with mild/moderate asthma. For this purpose, the investigators intend to evaluate the effect of a cold air exercise test on the Forced Expiratory Volume in 1 second (FEV1), respiratory symptoms, functional airway integrity, local and systemic inflammation and on the airway microbiome.

This study also features as an exploratory study for a subsequent interventional study in order to establish the feasibility of the cold air exercise protocol and to determine the extent of the effects in subjects with mild/moderate asthma.

DETAILED DESCRIPTION:
It is already demonstrated that exercising during cold air exposure and at a high altitude may induce asthmatic symptoms, a variable degree of airway obstruction and increased neutrophilic airway inflammation in asthmatic patients. Therefore, in this project, the investigators want to evaluate the feasibility, of a shorter standardized "cold air exercise test" (a submaximal exercise challenge in a controlled cold air (-5°C, relative humidity 60%) environment) and to compare the respiratory physiologic reactions to physical exercise during cold exposure between healthy volunteers and asthmatic patients. For this purpose, they intend to evaluate the effect of a cold air exercise test on FEV1, respiratory symptoms, functional airway integrity, local and systemic inflammation and on the airway microbiome.

This study features as an exploratory study for a subsequent interventional study, that will assess the protective effect of azithromycin versus placebo on the cold air exercise induced changes in patients with mild/moderate asthma (ALASCAIR2 study). The present preparatory study is needed to standardize the cold air exercise test in a controlled environment so that it would be possible to use it as challenge test in an interventional study and to identify the most appropriate design for such a study.

The primary objective of this study is to compare the proportional change in FEV1, pre to post a 90 minutes submaximal exercise in a cold air environment between healthy volunteers versus mild/moderate asthmatics, calculated as a time-weighted average over the 30 minutes post-exposure.

The primary endpoint is the change in FEV1, calculated as a time-weighted average over the 30 minutes after the cold exercise test. At each time point (pre-exposure, 5' post-exposure, and at 15, 25 and 35 minutes post-exposure), FEV1 (L) will be measured in triplicate.

They want to evaluate whether the exercise test in a cold air environment produces respiratory symptoms (such as nasal discharge or obstruction, dyspnea, cough and/or mucus production, etc.), has an impact on airway integrity (nasal patency, airflow obstruction, lung ventilation inhomogeneity & small airway dysfunction, bronchial hyperreactivity, cough reflex hypersensitivity), induces local or systemic inflammatory changes (biomarkers in nasal fluid, sputum and blood) or changes to the airway microbiome (in nasal fluid and sputum) in healthy volunteers and in mild/moderate asthmatics. The study group also want to compare the observed changes induced by the cold air exercise test between the healthy volunteers and the mild/moderate asthmatics.

The secondary endpoints of this study include the observed changes in (respiratory) symptom score, Peak Nasal Inspiratory Flow (PNIF), Forced Vital Capacity (FVC), Forced Expiratory Flow (FEF25-75), Fraction of Exhaled Nitric Oxide (FeNO), histamine provocative concentration causing 20% drop in FEV1 (PC20), cough threshold C2 & C5, sputum differential cell count, biomarkers in nasal fluid, sputum and blood, nasal and sputum microbial communities between the healthy volunteers and the mild/moderate asthmatics.

ELIGIBILITY:
INCLUSION CRITERIA - healthy volunteers

* age between 18 and 60 years at time of signing informed consent
* BMI between 18-28 kg/m2
* able to comply with study protocol, in the investigator's judgement
* non-smoking or ex-smokers for at least 12 months with less than 10 pack years
* no immunoglobulin E (IgE) mediated hypersensitivity
* normal spirometry & normal ECG at screening
* negative histamine provocation (defined as His- if PC20 >/= 8 mg/ml and His+ healthy controls if PC20 > 4 mg/ml and < 8 mg/ml)

INCLUSION CRITERIA - asthmatic patients

* age between 18 and 60 years at time of signing informed consent
* BMI between 18-28 kg/m2
* able to comply with study protocol, in the investigator's judgement
* non-smoking or ex-smokers for at least 12 months with less than 10 pack years
* physician-diagnosed asthma for more than 6 months
* post bronchodilator FEV1 of ≥ 80% at screening
* documented airway reversibility either by means of post bronchodilator reversibility of > 12% and > 200 ml or in the previous 6 months or by means of documented airway hyperresponsiveness (histamine PC20 <8 mg/ml) at screening
* Asthma Control Questionnaire (ACQ) < 1,5
* regular treatment with inhaled corticosteroids (ICS) with or without long-acting beta-agonists (LABA) (unchanged dose for at least 1 month)
* normal ECG at screening

EXCLUSION CRITERIA - healthy volunteers

* physician-diagnosed asthma or history of (post)infectious bronchial hyperreactivity
* major pulmonary or cardiovascular disease
* treatment with β-blockers
* pregnancy

EXCLUSION CRITERIA - asthmatics patients

* unable to produce sputum with sputum induction
* previous history of intubation or admission to the intensive care unit due to asthma
* severe asthma exacerbation within one year prior to screening visit
* treatment with oral or systemic steroids within one year prior to screening visit
* previous treatment with biologics for asthma
* treatment with β-blockers
* other major concurrent pulmonary (such as chronic obstructive pulmonary disease, cystic fibrosis, sarcoidosis, interstitial lung disease, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis, bronchiectasis) or cardiovascular disease
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 seconds (FEV1) | pre-, 5, 15, 25 and 35 minutes, 24 hours and 1 week post-exposure
  Change in FEV1, calculated as a time-weighted average over the 35 minutes after the cold air exercise test and 24 hours and 1 week post-exposure. A maximal fall of 10% will be considered as positive response

SECONDARY OUTCOMES:
Changes in asthma control | Pre-exposure and immediately, 24 hours and 1 week post-exposure
  Asthma control will be determined using the Asthma Control Questionnaire (ACQ-6), including 6 questions. Each question will be scored from 0-6 and added together. This final score will be divided by the number of questions. If ACQ-6 < 0.75 = controlled asthma, ACQ-6 from 0.75-1.5 = partly controlled asthma and ACQ-6 > 1.5 = uncontrolled asthma.
Changes in respiratory symptom score | Pre-exposure and immediately, 24 hours and 1 week post-exposure
  The degree of dyspnea will be determined using Borg scale. This Borg scale is 0 to 10 rated scale. With 0 no dyspnea and 10 complete dyspnea.
Cough hypersensitivity | Pre-exposure and 24 hours and 1 week post-exposure
  Cough hypersensitivity (Capsaicin cough threshold) will be measured using a capsaicin challenge test. The concentrations (µmol/l) which provokes 2 coughs (C2) and 10 coughs (C10) will be recorded and will be compared before and after cold air exposure.
Bronchial hyperreactivity | Pre-exposure and 1 week post-exposure
  Bronchial hyperreactivity will be measured using a histamine provocation. Bronchial hyperreactivity will be confirmed when there is a drop of 20% in FEV1 post histamine provocation (PC20).
Nasal hyperreactivity | Pre-exposure and immediately and 24 hours post-exposure
  Nasal hyperreactivity will be measured using a PNIF measurement. Nasal hyperreactivity will be confirmed when there is a drop of 20% in PNIF.
Airway inflammation | Pre-exposure and 24 hours and 1 week post-exposure
  Bronchial airway inflammation. Differential cell count will be performed on sputum samples, determining eosinophilic (>3% eosinophils, <61% neutrophils), neutrophilic (<3% eosinophils and >61% neutrophils), pauci-granulocytic (<3% eosinophils and <61% neutrophils) and mixed granulocytic airway inflammation (>3% eosinophils and >61% neutrophils).
Cytokine pattern in the airways | Pre-exposure and 24 hours and 1 week post-exposure
  Cytokines concentrations (pg/ml) will also be determined in sputum supernatant using a U-plex assay.
Biomarkers for airway inflammation | Pre-exposure and 24 hours and 1 week post-exposure
  FeNO will be used as biomarker for eosinophilic airway inflammation. FeNO < 25 ppb = eosinophilic inflammation less likely, FeNO between 25 and 50 ppm = need further interpretation with additional clinical information, FeNO > 50 ppm = indication of eosinophilic airway inflammation (according to the American Thoracic Society guidelines)
Nasal inflammation | Pre-exposure and immediately and 24 hours post-exposure
  Cytokine concentrations (pg/ml) will be determined in the nasal fluid as biomarkers for nasal inflammation
Systemic inflammation | Pre-exposure and immediately, 24 hours and 1 week post-exposure
  The degree of system inflammation will be determined via differential blood cell count.
Biomarkers for systemic inflammation | Pre-exposure and immediately, 24 hours and 1 week post-exposure
  The degree of system inflammation will be determined via C-reactive protein (CRP) levels. Normal values for CRP are considered < 10 mg/ml.
Changes in microbiome in lung and nose | Pre-exposure and 1 week post-exposure
  The presence of 22 common respiratory viruses, 5 bacteria and 1 fungi will be determined using qualitative reverse transcription polymerase chain reaction (qRT-PCR) in sputum and nasal fluid. Pre and post-exposure microbiome patterns will be compared.
Evaluation of the heart rate pattern | Pre-exposure and during the 90 minutes cold air exposure
  Cardiovascular health will be evaluated by determining the heart rate pattern using ECG. Deviation from a normal ECG pattern will be recorded.
Determining the exercise capacity | Pre-exposure
  Exercise capacity will be checked. In a single test pre-exposure, the aerobic heart rate zone, anaerobic heart rate zone and maximal oxygen volume uptake (VO2max) heart rate zone will be evaluated to determine the exercise capacity

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Dupont, Prof. dr, Principal Investigator — KU Leuven/ UZ Leuven
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No